CLINICAL TRIAL: NCT06898294
Title: Assessment of Kidney Function by Self-administrable and Portable Electrical Impedance Tomography (EIT)
Brief Title: Assessment of Kidney Function by Electrical Impedance Tomography (EIT)
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Desmond Yat-Hin Yap, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: HKU-YAP-EIT-KF01
Record Dates: First submitted 2024-12-13; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: Electrical Impedance Tomography; Kidney Function Assessment; Biomedical Imaging
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patient's blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with chronic kidney disease: Adults who are clinically diagnosed with CKD at different stages (stage 1-5).
  Interventions: Diagnostic Test: EIT kidney function assessment
- Healthy volunteers (controls): Healthy adults who do not have any known kidney diseases will be examined
  Interventions: Diagnostic Test: EIT kidney function assessment

INTERVENTIONS:
Diagnostic Test: EIT kidney function assessment — The product under investigation is named Gense EIT-kidney device. This kidney device is a portable and non-invasive imaging modality capable of capturing the cross-sectional bioelectrical impedance distribution of the kidney at multiple current injection frequencies using electrical impedance tomography (EIT). Currently, the kidney device employs a band consisting of 16 equally distributed electrodes around the abdomen. The electrode band is connected to a control unit that switches the electrode stimulation and measurement pairs, then sends the collected measurement to a computational unit for image reconstruction. The images are then post-processed to extract functional kidney images for diagnosis. This kidney device has a large LED screen, allowing the functional images to be produced and visualized.

SUMMARY:
The product under investigation is named Gense EIT-kidney device. This kidney device is a portable and non-invasive imaging modality capable of capturing the cross-sectional bioelectrical impedance distribution of the kidney at multiple current injection frequencies using electrical impedance tomography (EIT). Currently, the kidney device employs a band consisting of 16 equally distributed electrodes around the abdomen. The electrode band is connected to a control unit that switches the electrode stimulation and measurement pairs, then sends the collected measurement to a computational unit for image reconstruction. The images are then post-processed to extract functional kidney images for diagnosis. This kidney device can connect to an external screen, allowing the functional images to be produced and visualized.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is an escalating health problem in the global and local perspective. CKD is defined as all disorders affecting kidney structures and functions. The main classifications are acute kidney injury (AKI) for kidney diseases where symptoms last within one week and CKD where the renal abnormalities last for more than 3 months. AKI and CKD are interrelated; AKI can progress into CKD, and CKD can further progress and comorbid with hypertension, diabetes, and cardiovascular diseases. Based on the 2012 KDIGO (Kidney Disease: Improving Global Outcomes) guidelines, the criteria for CKD diagnosis relies on functional measurements based on the glomerular filtration rate (GFR), while the structural markers of kidney damage are assessed with imaging technique such as renal ultrasound. CKD can classified into five stages (Stage 1: Normal/ high function; Stage 2: Mildly decreased function; Stage 3: Mild to moderately decreased function; Stage 4: Severely decreased function; Stage 5: Kidney failure) based on the GFR. The last stage is referred to as end-stage renal disease (ESRD) that the patient requires dialysis support or a kidney transplant. Unlike most diseases, symptoms of most kidney problems are non-specific, and patients are often asymptomatic until advanced stages. It is estimated that 90% of those with CKD are not aware of their condition. According to the Department of Health of HKSAR, there were 21.3 million incident cases, 1.2 million deaths and 35 million years of disability-adjusted like years (DALYs) globally in 2016, an 88.8%, 98% and 62.2% increase from 1990, respectively. Recent analysis suggests that the age-standardised global prevalence of CKD was greater in women than men. However, the rate of progression into ESRD and risk of mortality are significantly more pronounced in men compared to women, except in post-menopausal and diabetic female patients. Furthermore, seniors older than 60 years of age are major risk groups for CKD as the risk of diabetes mellitus and high blood pressure increases with age.

The gold standard of kidney function assessment to diagnose and classify CKD stages is measuring the GFR in patients. The stages of CKD can be classified as follows: Stage 1 is kidney damage with normal or increased GFR (>90 mL/min); Stage 2 is a mild reduction in GFR (60-89 mL/min); Stage 3 is a moderate reduction in GFR, in which Stage 3a (45-59 mL/min) and Stage 3b (30-44 mL/min); Stage 4 is a severe reduction in GFR (15-29 mL/min); Stage 5 is kidney failure or ESKD in which GFR < 15 mL/min or dialysis is facilitated. The gold standard of kidney function assessment to diagnose CKD is the direct measurement of GFR over 24 hours urine collection, but this is impractical. The alternative methods are measured GFR (mGFR), which measures clearance of exogenous markers such as inulin, iohexol, and iothalamate, and estimated GFR (eGFR) based on endogenous filtration markers, serum creatinine and urea, though none can precisely represent the true GFR. Exogenous markers, specifically urinary inulin clearance, is considered superior to measure GFR, but they are labour-intensive procedures and too expensive for repeated use. In clinical settings, the conventional method is the usage of estimated equations to measure eGFR in lieu of mGFR for its simplicity and speed. However, it was observed that eGFR equations are susceptible to overestimation of kidney function in physically weak patients, for example the elderly individuals. Thus, this method only serves as the best estimate of GFR levels and it does not represent the true GFR. Furthermore, currently there is no standardization for the range of mGFR measurements used as the basis for estimated equations, which is why this approach is doubted for biases and inaccuracy.

Since the biochemical measurements might be inadequate for kidney function assessment, as these tests are insensitive and not able to discriminate the causes of kidney diseases though some of them have different functional consequences. Imaging modalities, such as ultrasound (US) and computed tomography (CT), are increasingly employed to improve the diagnosis of kidney diseases, as well as reveal morphological changes in kidney structure and composition. However, US shows limited ability to identify increased cortical echogenicity caused by chronic kidney failure, thereby making it difficult to rule out the reversible causes of renal failure. As for CT, the application of intravenous iodinated contrast leads to its contraindication in advanced renal failure, while the presence of ionizing radiation leads to its contraindication in early pregnancy cases. The discharge of potentially toxic contrast agent is limited to patients show an estimated glomerular filtration rate (eGFR) under 30 ml/minute.

Further, renal biopsy with invasive extraction of kidney tissue for histological analysis could identify the type and severity of the kidney disease. Biopsy can be used to reveal scarring, inflammation and protein deposit which are unrecognizable with ultrasound, blood, and urine tests. However, percutaneous biopsy guided by imaging modalities or open biopsy which employs surgical methods, making it more invasive and exposing the risks of post-procedure lesion and infection to both targeted and nearby areas.

Here, EIT could be an alternative low cost, accessible, ionizing radiation-free and contrast agent-free non-invasive imaging technique to detect both structural and functional changes within the kidney. Gense EIT-Kidney scan is quick (~10 minutes), portable and does not require a trained operator. Existing EIT commercial devices are at present being deployed in some clinical settings. EIT technology has been in use since more than a decade, although so far it has mostly been used to assist mechanically ventilated patients in intensive care units to prevent lung damage caused by artificial ventilation. Dräger's EIT lung imaging device (PulmoVista® 500) has been shown to detect the regional distribution of ventilation in real-time and guide mechanical ventilation changes, including assessing the optimal PEEP and pulmonary compliance. Another commercial EIT device is Enlight® (Timpel, Brasil), which can also assist in early identification of patient-ventilator dyssynchrony and continuously quantify regional pulmonary ventilation heterogeneity.

Within the past few years, several exploratory studies have been performed on applying bioelectrical impedance in assisting kidney function assessment in animal models such as pigs. Impedance measurements have also applied on improving the estimation of GFR in chronic kidney disease patients. The electrical conductivity of biological tissues varies according to the tissue type and frequency of AC current. On the other hand, kidney tissue conductivity significantly increases over frequency change. Hence, biological tissues can potentially be differentiated using EIT frequency spectrum analysis.

For kidney function assessment, GFR remains a good measure. However, its limitations need to be addressed. The core limitation is that estimated equations as the clinical standard to measure eGFR is meant to calibrate differences in muscle mass, which is the source of serum creatinine, based on demographic variables such as age, sex, gender, race, etc, but it still does not account for individual variability in muscle mass. EIT could be the alternative to predict GFR based on the body bioelectrical impedance, which correlated appendicular lean mass (ALM) for skeletal muscle mass calculation, which previously demonstrated by bioelectrical impedance analysis with resistance and reactance. Not only does this method potentially give a more accurate estimate of GFR, but it also gives a good prediction of the functional capacity, quality of life and outcome in CKD.

The aim of this study is to verify and validate the relation between EIT and GFR measurements for functional analysis of the kidneys. This study will also study the feasibility of EIT as a potential imaging modality to analyse the structure problems in the patients with kidney disease. GFR based on equations with bioelectrical impedance involvement will be compared to GFR based on urinary inulin clearance as the gold standard. Finally, demographics, clinical assessment and patient history will be considered for further analysis. The results from this project will develop EIT as a convenient and non-invasive screening test for kidney dysfunction and CKD. The early detection of CKD will enable timely interventions to retard further deterioration of renal function and thus improve overall patient outcomes and healthcare resource utilizations.

ELIGIBILITY:
Inclusion Criteria:

- clinically diagnosed with CKD at different stages (stage 1-5) of the disease based on GFR measurement results Age: 18-90. Gender: Male/ Female

Exclusion Criteria:

* ● Subjects with known kidney disease or abnormalities (for the control group).

  * Subjects who had any kind of kidney surgery or kidney transplantation.
  * Subjects with damaged skin on the abdomen.
  * Subjects with implanted electronic devices.
  * Subjects with spinal diseases/discomfort
  * Subjects who had any recent abdominal surgery
  * Pregnant women.
  * Obese subjects (BMI>35).
  * Subjects with uncontrollable involuntary body movements such as degenerative disorders (e.g., Alzheimer's and Parkinson's disease); Seizure disorders (e.g., epilepsy, stroke, neuroleptic drugs); Neurological disorders (e.g., tardive dyskinesia and cerebral palsy, tremors, myoclonus, tics, athetosis, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kidney disease subjects Patients between the age group of 18-90, clinically diagnosed with CKD at different stages (stage 1-5) of the disease based on GFR measurement results, between the age group of 18-90 will be included.
  Healthy volunteers (Controls) In this group, healthy adults who do not have any known kidney diseases will be examined. Healthy subjects will be chosen to be age and gender-matched with case subjects. Healthy volunteers will have blood and urine tests to confirm that they have normal renal function.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Identification of optimal EIT current injection frequencies for kidney function assessment | 6 months
  Multiple current injection frequencies ranging from 10kHz to 350kHz will be used and corresponding EIT images will be reconstructed based on frequency difference based relative EIT imaging. The optimal range of stimulation frequency will be identified based on multiple factors, including: image reconstruction repeatability and reproducibility, signal to noise ratio (SNR), consistency between expected tissue responses and imaging results. investigations will be performed to identify optimal frequency ranges for the assessment of kidney function.
Functional assessment comparison between GFR measurement and EIT-Kidney scanning | 12 months
  Recruited subjects will be classified into five different kidney functional stages (Stage 1-5) according to existing classification standard. Subjects will undergo GFR measurements and EIT imaging. It is preferred that both EIT and GFR measurements are conducted separately. Kidney function test results between GFR measurements and EIT will be performed in order to identify the feasibility and accuracy of EIT-kidney device. Common kidney functional indicator (e.g., EIT predicted GFR) would also be derived from continuous EIT functional images.
Demographics, clinical assessments, and patient history analysis | 6 months
  The EIT-derived indicators will be analyzed together with demographics, clinical assessments and patient history to derive fine grained insights and elucidate the effect of demographics and biometrics on EIT kidney data. The parameters include, but not limited to, age, chest size, gender, weight, height, BML, smoking habits and ethnicity. The analysis will improve the stability of the EIT indicators, and ultimately increase their predictive power towards diseased kidney regions.

CONTACTS AND LOCATIONS:
Overall Officials: Yat Hin, Desmond Yap, PhD, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunne E, OHalloran M, Craven D, Puri P, Frehill P, Loughney S, Porter E. Detection of Vesicoureteral Reflux Using Electrical Impedance Tomography. IEEE Trans Biomed Eng. 2019 Aug;66(8):2279-2286. doi: 10.1109/TBME.2018.2886830. Epub 2018 Dec 14. PMID 30571612
- [Background] Chen X, Kao TJ, Ashe JM, Boverman G, Sabatini JE, Davenport DM. Multi-channel electrical impedance tomography for regional tissue hydration monitoring. Physiol Meas. 2014 Jun;35(6):1137-47. doi: 10.1088/0967-3334/35/6/1137. Epub 2014 May 20. PMID 24845597
- [Background] Macdonald JH, Marcora SM, Jibani M, Roberts G, Kumwenda MJ, Glover R, Barron J, Lemmey AB. Bioelectrical impedance can be used to predict muscle mass and hence improve estimation of glomerular filtration rate in non-diabetic patients with chronic kidney disease. Nephrol Dial Transplant. 2006 Dec;21(12):3481-7. doi: 10.1093/ndt/gfl432. Epub 2006 Sep 5. PMID 16954169
- [Background] You F, Shi X, Shuai W, Zhang H, Zhang W, Fu F, Liu R, Xu C, Bao T, Dong X. Applying electrical impedance tomography to dynamically monitor retroperitoneal bleeding in a renal trauma patient. Intensive Care Med. 2013 Jun;39(6):1159-60. doi: 10.1007/s00134-013-2895-y. Epub 2013 Mar 29. No abstract available. PMID 23539146